CLINICAL TRIAL: NCT01411020
Title: Target-controlled Infusion (TCI) of Propofol for Induction in Children 3 to 11 Years
Brief Title: Target-controlled Infusion of Propofol for Induction of Pediatric Anesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Principal Investigator, Ricardo Fuentes Henriquez, Profesor Asistente, Departamento de Anestesiología, Pontificia Universidad Catolica de Chile
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ricardo Fuentes; Hernan Muñoz
Record Dates: First submitted 2011-08-03; First posted 2011-08-05 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2009-08

CONDITIONS: Children Under General Anesthesia
MeSH Terms: interventions — Intubation, Intratracheal

ARMS (10):
- Grupo 1 (Experimental): Doses of induction: propofol 4 mcg/ml and fentanyl 3 mcg/kg
  Interventions: Procedure: endotracheal intubation
- Grupo 2 (Experimental): Dose of induction: propofol 4.5 mcg/ml and fentanyl 3 mcg/kg
  Interventions: Procedure: endotracheal intubation
- Grupo 3 (Experimental): Doses of propofol: propofol 5 mcg/ml and fentanyl 3 mcg/kg
  Interventions: Procedure: endotracheal intubation
- Grupo 4 (Experimental): Doses of induction: propofol 5.5 mcg/ml and fentanyl 3 mcg/kg
  Interventions: Procedure: endotracheal intubation
- Grupo 5 (Experimental): Doses of induction: propofol 6 mcg/ml and fentanyl 3 mcg/kg
  Interventions: Procedure: endotracheal intubation
- Grupo 6 (Experimental): Doses of induction: propofol 4 mcg/ml and fentanyl 5 mcg/kg
  Interventions: Procedure: endotracheal intubation
- Grupo 7 (Experimental): Doses of induction: propofol 4.5 mcg/ml and fentanyl 5 mcg/kg
  Interventions: Procedure: endotracheal intubation
- Grupo 8 (Experimental): Doses of induction: propofol 5 mcg/ml and fentanyl 5 mcg/kg
  Interventions: Procedure: endotracheal intubation
- Grupo 9 (Experimental): Doses of induction: propofol 5.5 mcg/ml and fentanyl 5 mcg/kg
  Interventions: Procedure: endotracheal intubation
- Grupo 10 (Experimental): Doses of induction: propofol 6 mcg/ml and fentanyl 5 mcg/kg
  Interventions: Procedure: endotracheal intubation

INTERVENTIONS:
Procedure: endotracheal intubation — to perform endotracheal intubation if number of bispectral index (BIS) is 40-60,

SUMMARY:
The purpose of this study is to determine a effect-site concentration of propofol in children 3 to 11 years effective to make a induction of general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* obtained informed consent
* children between 3 and 11 years
* healthy
* elective surgery under general anesthesia
* no premedication

Exclusion Criteria:

* body mass index for age > 95th percentile
* chronic or acute intake of any sedative drug
* any known adverse effect to the study drugs

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2009-10; Primary Completion 2012-08 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
dose of propofol | two days (duration of hospitalization)
  to obtain a dose appropriate of propofol in induction of anesthesia

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinico Universidad Catolica, Santiago, Santiago Metropolitan, Chile

REFERENCES:
- [Background] Munoz HR, Leon PJ, Fuentes RS, Echevarria GC, Cortinez LI. Prospective evaluation of the time to peak effect of propofol to target the effect site in children. Acta Anaesthesiol Scand. 2009 Aug;53(7):883-90. doi: 10.1111/j.1399-6576.2009.01995.x. Epub 2009 Jun 3. PMID 19496767